CLINICAL TRIAL: NCT01123096
Title: Is the Cough Stress Test Equivalent to the 24 Hour Pad Test in the Assessment of Stress Incontinence?
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Karen Noblett, Division Director, University of California, Irvine
Other Study IDs: 2007-5923
Record Dates: First submitted 2010-05-06; First posted 2010-05-14 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stress Urinary Incontinence: Patients with the primary complaint of stress incontinence with minimal or no urge incontinence symptoms. They must be able to read English as the study involves use of validated questionnaires which have only been validated in English.
  Interventions: Procedure: Cough Stress Test; Other: 24 Hour Pad Test

INTERVENTIONS:
Procedure: Cough Stress Test — A cough stress test is performed by using a catheter to introduce 300ml of sterile water into the bladder. The patient is then asked to stand and cough forcefully and the clinician will observe for urine loss.
Other: 24 Hour Pad Test — The patient will be provided with a standard number of pads in a sealed bag that have been pre-weighed. The patient will wear the pads for 24 consecutive hours then return the all the pads within the bag for weighing post usage.

SUMMARY:
The purpose of this research study is to identify if the cough stress test is equal to the 24hour pad test in assessing stress urinary incontinence.

DETAILED DESCRIPTION:
The 24 hour pad test involves women collecting their pre-weighed incontinence pads for 24 hours and returning them to the clinician for weighing. This allows for accurate quantification of urine loss. This test is often used in clinical studies before and after intervention to assess efficacy of treatment.

The cough stress test is an alternative testing modality used to evaluate stress incontinence. It is an easy test to perform in a single visit to the clinician's office and the results are immediately available. It involves the patient coughing forcefully with a full bladder and watching for leakage of urine through the urethra.

In our study, our primary aim is to compare the equivalency of the cough stress test to the 24 hour pad test as a measure of stress urinary incontinence. Our secondary aim will be to assess patient comfort and satisfaction with each of the testing modalities. If the cough stress test is equivalent, it will provide an additional, easy to use tool for patient evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients with the primary complaint of stress incontinence with minimal or no urge incontinence symptoms. They must be able to read English as the study involves use of validated questionnaires which have only been validated in English.

Exclusion Criteria:

* patients unable to stand (to perform standing stress test), patients with leakage from a urinary tract fistula, use of vaginal creams within 72 hours of the pad test, active vaginal infection, sexual intercourse within 24 hours of the pad test and patients who do not read English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the primary complaint of stress incontinence with minimal or no urge incontinence symptoms. They must be able to read English as the study involves use of validated questionnaires which have only been validated in English.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary aim is to compare the equivalency of the cough stress test to the 24 hour pad test as a measure of stress urinary incontinence. | Data will be analyzed at study completion at approximately 3 years.

SECONDARY OUTCOMES:
The secondary aim will be to assess patient comfort and satisfaction with each of the testing modalities. If the cough stress test is equivalent, it will provide an additional, easy to use tool for patient evaluation. | Data will be analyzed at study completion at approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Noblett, MD, Principal Investigator — UCI Medical Center
Locations (1):
- UC Irvine Women's Healthcare, Orange, California, United States